CLINICAL TRIAL: NCT02659189
Title: Hospitalary Chronic Obstructive Pulmonary Disease Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 2677
Record Dates: First submitted 2016-01-05; First posted 2016-01-20 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: COPD Exacerbations; Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create an institutional registry of Chronic Obstructive Pulmonary disease through a prospective survey based on epidemiological data, risk factors, diagnosis, prognosis, treatment, monitoring and survival.

DETAILED DESCRIPTION:
The main goal is to describe the characteristics of chronic obstructive pulmonary disease patients, including their clinical, spirometric, exacerbation and mortality characteristics within the population of the Hospital Italiano de Buenos Aires.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years with a chronic obstructive pulmonary disease diagnosis according to global obstructive lung Global initiative for chronic Obstructive Lung Disease criteria.
* Follow up at the Hospital Italiano de Buenos Aires.

Exclusion Criteria:

* Refusal to participate or to agree to the informed consent.
* Known non chronic obstructive pulmonary disease respiratory disease (ej: Lung Cancer, Tuberculosis, Pulmonary Fibrosis, Neumoconiosis, Cystic Fibrosis, Sarcoidosis, etc)
* Severe alpha-1 antitripsin deficit (typr SZ or ZZ)
* Previously thoracic surgery (ej: lung volume reduction, lung transplantation).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 40 years with a chronic obstructive pulmonary disease diagnosis according to global initiative for chronic obstructive lung disease criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Death | At 6 months after enrollment
  All cause of death

SECONDARY OUTCOMES:
Morbidity | At 6 months after enrollment
  Saint George respiratory questionnaire
Functional decline (Forced expired volume at one second) | At 12 months after enrollment
  Forced expired volume at one second
Exacerbations (defined as an increase in symptoms that requires treatment) | At 12 months after enrollment
  Number of exacerbations in the timeframe (defined as an increase in symptoms that requires treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muiño Adriana, María Victoria López Varela, and Ana María Menezes. Prevalencia de la enfermedad pulmonar obstructiva crónica y sus principales factores de riesgo: proyecto platino en Montevideo. Revista Médica del Uruguay. 2005;21: 37-48
- [Background] Moreira GL, Gazzotti MR, Manzano BM, Nascimento O, Perez-Padilla R, Menezes AM, Jardim JR. Incidence of chronic obstructive pulmonary disease based on three spirometric diagnostic criteria in Sao Paulo, Brazil: a nine-year follow-up since the PLATINO prevalence study. Sao Paulo Med J. 2015 May-Jun;133(3):245-51. doi: 10.1590/1516-3180.2015.9620902. Epub 2015 Jun 1. PMID 26176929